CLINICAL TRIAL: NCT03547024
Title: An Open-Label Drug Interaction Study in Healthy Subjects to Evaluate the Effects of Multiple Doses of JNJ55308942 on the Cytochrome P450 CYP3A4, CYP2D6 and CYP2C19 Activity and on the Pharmacokinetics of Levonorgestrel/Ethinyl Estradiol
Brief Title: A Study in Healthy Participants to Evaluate the Effects of Multiple Doses of JNJ-55308942 on Cytochrome P450 Substrate Activity and on the Pharmacokinetics of Levonorgestrel/Ethinyl Estradiol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108486; 2018-000194-75 (EudraCT Number); 55308942EDI1003 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-55308942; Levonorgestrel; Ethinyl Estradiol; Omeprazole; Dextromethorphan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: JNJ-55308942 + Drug Cocktail (Experimental): Participants will receive a single dose of drug cocktail on Day 1 followed by JNJ-55308942 high dose once daily from Day 3 to Day 14 and a single dose of drug cocktail on Day 12.
  Interventions: Drug: JNJ-55308942 High Dose; Drug: Drug Cocktail:Midazolam (2mg)/Omeprazole (20mg)/Dextromethorphan (30mg)
- Part 2: JNJ-55308942 + Levonorgestrel/Ethinyl Estradiol (Experimental): Participants will receive a single dose of levonorgestrel/ethinyl estradiol alone on Day 1 followed by JNJ-55308942 high dose once daily on Days 5 to 18 and a single dose of levonorgestrel/ethinyl estradiol on Day 14.
  Interventions: Drug: JNJ-55308942 High Dose; Drug: Levonorgestrel/Ethinyl Estradiol Fixed Dose combination (FDC); Drug: Drug Cocktail:Midazolam (2mg)/Omeprazole (20mg)/Dextromethorphan (30mg)
- Part 3: JNJ-55308942 + Drug Cocktail (Experimental): Participants will receive a single dose of drug cocktail alone on Day 1 followed by JNJ-55308942 low dose once daily on Days 3 to Day 14 and a single dose drug cocktail on Day 12.
  Interventions: Drug: JNJ-55308942 Low Dose; Drug: Drug Cocktail:Midazolam (2mg)/Omeprazole (20mg)/Dextromethorphan (30mg)

INTERVENTIONS:
Drug: JNJ-55308942 High Dose — Participants will receive high dose of JNJ-55308942 orally once daily.
  Arms: Part 1: JNJ-55308942 + Drug Cocktail; Part 2: JNJ-55308942 + Levonorgestrel/Ethinyl Estradiol
Drug: JNJ-55308942 Low Dose — Participants will receive low dose of JNJ-55308942 orally once daily.
  Arms: Part 3: JNJ-55308942 + Drug Cocktail
Drug: Levonorgestrel/Ethinyl Estradiol Fixed Dose combination (FDC) — Participants will receive 0.150 milligram (mg) levonorgestrel and 0.030 mg ethinyl estradiol FDC tablet orally.
  Other Names: Microgynon 30
  Arms: Part 2: JNJ-55308942 + Levonorgestrel/Ethinyl Estradiol
Drug: Drug Cocktail:Midazolam (2mg)/Omeprazole (20mg)/Dextromethorphan (30mg) — Participants will receive single dose of drug cocktail consisting of midazolam (2 mg), dextromethorphan (30mg) and omeprazole (20 mg) orally.

SUMMARY:
The purpose of this study is to determine the effect of JNJ-55308942: 1) high dose at steady state on the single dose pharmacokinetics of a cocktail containing selective probes of cytochrome P450 (CYP) enzymes (CYP3A, CYP2D6 and CYP2C19) in healthy adult participants (Part 1); 2) high dose at steady state on the single dose pharmacokinetics of a combination oral contraceptive containing levonorgestrel and ethinyl estradiol in healthy female participants (Part 2); and 3) low dose at steady state on the single dose pharmacokinetics of a cocktail containing selective probes of CYP enzymes (CYP3A, CYP2D6 and CYP2C19) in healthy adult participants (Part 3).

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2), inclusive (BMI = weight/height^2)
* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and first admission (Day -1) to the clinical unit. Minor abnormalities in ECG, which are not considered to be of clinical significance by the physician investigator, are acceptable
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel [excluding liver function tests], hematology [including coagulation], or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities to be not clinically significant. This determination must be recorded in the participant's source documents and initialed/signed by the physician investigator
* All women of child-bearing potential must have a negative highly sensitive serum (beta human chorionic gonadotropin [beta hCG]) at screening and a negative urine pregnancy test on Day -1
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 1 month after the last study drug administration

Exclusion Criteria:

* History of or current liver or renal insufficiency; significant skin disease such as, but not limited to, dermatitis, eczema, Stevens-Johnson Syndrome, drug rash, psoriasis or urticaria, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic (including coagulation disorders), rheumatologic, psychiatric, or metabolic disturbances, any inflammatory illness or any other illness that the Investigator considers should exclude the participant
* History of or current positive testing for hepatitis B surface antigen (HBsAg), Hepatitis B core (HBcAb) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening
* History of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that, in the opinion of the investigator, with written concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence)
* History of at least drug or alcohol use disorder according to Diagnostic and Statistical Manual of Mental Disorders (latest edition DSM-5) criteria within 6 months before screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Parts 1 and 3: Maximum Observed Analyte Concentration (Cmax) of Each Probe Substrate in Cocktail | Predose, 15 minute (min), 30min, 45min, 1 hour (h), 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 18h on Days 1 and 12
  Cmax of probe substrates in cocktail containing selective probes of CYP enzymes (CYP3A, CYP2D6 and CYP2C19) will be determined.
Parts 1 and 3: Area Under the Analyte Concentration-Time Curve from Time Zero to the Time of the Last Measurable Concentration (AUC[0-last]) of Each Probe Substrate in Cocktail | Predose, 15min, 30min, 45min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 18h on Days 1 and 12
  AUC(0-last) of probe substrates in cocktail containing selective probes of CYP enzymes (CYP3A, CYP2D6 and CYP2C19) will be determined.
Parts 1 and 3: Area Under the Analyte Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Each Probe Substrate in Cocktail | Predose, 15min, 30min, 45min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 18h on Days 1 and 12
  AUC (0-infinity) of probe substrates in cocktail containing selective probes of CYP enzymes (CYP3A, CYP2D6 and CYP2C19) will be determined.
Part 2: Cmax of Levonorgestrel and Ethinyl Estradiol | Predose, 15min, 30min, 45min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 18h on Days 1 and 14
  Cmax is the maximum observed analyte concentration.
Part 2: AUC(0-last) of Levonorgestrel and Ethinyl Estradiol | Predose, 15min, 30min, 45min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 18h on Days 1 and 14
  AUC(0-last) is defined as the area under the analyte concentration-time curve from time 0 to time of the last quantifiable concentration.
Part 2: AUC(0-infinity) of Levonorgestrel and Ethinyl Estradiol | Predose, 15min, 30min, 45min, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 18h on Days 1 and 14
  AUC (0-infinity) is the area under the analyte concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the analyte concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Parts 1, 2 and 3: Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability | Approximately 10 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Parts 1, 2 and 3: Observed Analyte Concentration Just Prior to the Beginning or at the end of a Dosing Interval (Ctrough) of JNJ-55308942 | Predose on Days 4 to 11, predose, up to 72 hours postdose on Day 12 (Parts 1 and 3); Predose on Days 5 to 13, predose, up to 120 hour postdose on Day 14 (Part 2)
  Ctrough is the observed analyte concentration just prior to the beginning or at the end of a dosing interval in a multiple dosing regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium